CLINICAL TRIAL: NCT02362113
Title: Glycemic Index, Glycemic Load and Common Psychological Disorders
Brief Title: Glycemic Index/ Load and Mental Disorders
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Leila Azadbakht, Department of Community Nutrition, School of Nutrition and Food Science, Isfahan University of Medical Sciences
Other Study IDs: 1364
Record Dates: First submitted 2015-02-02; First posted 2015-02-12 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Depression; Anxiety; Psychological Distress
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Isfahani adults: GI/GL
  Interventions: Other: GI/GL

INTERVENTIONS:
Other: GI/GL — GI and GL would be categorized as tertile. due to cross-sectional design of this study, intervention would not be applicable.

SUMMARY:
A total of 300 adults would be included in the present cross-sectional study. glycemic index (GI) and glycemic load (GL) would be assessed by using a validated self-administered dish-based semi-quantitative food frequency questionnaire. Validated Iranian versions of Hospital Anxiety and Depression Scale and General Health Questionnaire-12 would be used to assess anxiety, depression and psychological distress.

DETAILED DESCRIPTION:
Frequency of 5 food groups will be asked in dish-based semi-quantitative food frequency questionnaire and they would be converted to grams. GI and GL will be estimated by using international table of GI and GL.

Validated Iranian versions of Hospital Anxiety and Depression Scale and General Health Questionnaire (GHQ)-12 were used to assess anxiety, depression and psychological distress.

Possible score range for anxiety and depression is from 0 to 21. Scores of 8 or higher on either section were considered as the presence of anxiety or depression and scores of 7 or less were considered as normal status. In the present study, participants who got scores of 4 or more from GHQ were considered to have psychological distress.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-75 years of free-living individuals.

Exclusion Criteria:

* Over or underestimating of total energy intake
* Uncompleted questionnaire (more than 30% of questions)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: non-academic staff of Isfahan University of Medical Sciences (IUMS), Isfahan, Iran, who were working in hospitals, university campus and health centers affiliated with IUMS
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-04 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
odds ratio for having depression resulted from statistical analysis | up to 4 months

SECONDARY OUTCOMES:
depression score resulted from Hospital Anxiety and Depression Scale | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Peyman Adibi, MD, Study Chair — Integrative Functional Gastroenterology Research Center, Isfahan University of Medical Sciences, Isfahan, Iran

REFERENCES:
- [Derived] Haghighatdoost F, Azadbakht L, Keshteli AH, Feinle-Bisset C, Daghaghzadeh H, Afshar H, Feizi A, Esmaillzadeh A, Adibi P. Glycemic index, glycemic load, and common psychological disorders. Am J Clin Nutr. 2016 Jan;103(1):201-9. doi: 10.3945/ajcn.114.105445. Epub 2015 Nov 25. PMID 26607943